CLINICAL TRIAL: NCT04850183
Title: Effect of Education on Disease Management to Women With Rheumatoid Arthritis on the Quality of Life and Levels of Anxiety and Depression
Brief Title: Effect of Education in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Irem Yildiz Cilengiroglu, Principal Investigator, Trakya University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/02
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis; Quality of Life; Depression, Anxiety; Nurse's Role
MeSH Terms: conditions — Arthritis, Rheumatoid; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients were interviewed twice, at baseline and at the 3rd month. All forms were applied to the patients in the intervention group at baseline. The patients were assigned to the intervention group at random and participated in a one-to-one training program consisting of a 30-min onset session. The Rheumatoid Arthritis Patient Education Booklet prepared by the researchers was administered to patients in the intervention group during education. In the 3rd month, all forms were applied again to the patients in the intervention group.
  Interventions: Behavioral: Education on disease management on the quality of life, and anxiety and depression about Rheumatoid Arthritis
- Control group (No Intervention): Patients were interviewed twice, at baseline and at the 3rd month. All forms were applied to the patients in the control group at baseline. In the 3rd month, the same forms were applied to the untrained patients in the control group.

INTERVENTIONS:
Behavioral: Education on disease management on the quality of life, and anxiety and depression about Rheumatoid Arthritis — The patients in the intervention group participated in a one-to-one training program consisting of a 30-min onset session.
  Arms: Intervention group

SUMMARY:
This randomized controlled study aimed to determine the effect of education on disease management on the quality of life, and anxiety and depression levels of women with Rheumatoid Arthritis.

The hypotheses of the current study are as below:

H0: Education on disease management in women with Rheumatoid Arthritis does not affect the quality of life and anxiety and depression levels.

H1: Education on disease management in women with Rheumatoid Arthritis affects the quality of life and anxiety and depression levels.

Patients and Methods: The study was conducted with 66 women with Rheumatoid Arthritis (32 intervention, 34 control groups) at the rheumatology clinic and polyclinic of a university hospital between February and October 2019, in the city of Edirne, Turkey. Data were collected with "Patient Information Form", "Rheumatoid Arthritis Quality of Life Scale", "Health Assessment Questionnaire" and "Hospital Anxiety Depression Scale".

DETAILED DESCRIPTION:
Study design and participants This pretest and posttest prospective study was conducted as randomized controlled between February 2019 and October 2019 in the outpatient and inpatient clinics of the Department of Rheumatology of a university hospital in Edirne, Turkey.

Two study groups, control (n = 40) and intervention (n = 40) were randomized controlled groups with 80% power analysis and 95% confidence interval. A single-blind technique was used to eliminate any bias. The patients were not informed of the group to which they belonged. The patients were selected using a simple random sampling method and divided into intervention and control groups using the Research Randomizer program. In the intervention group, 40 women with RA were interviewed at baseline (first interview). In the 3rd month (last interview), eight patients were excluded for the following reasons: four did not wish to continue the study, three could not be reached, and one patient did not complete the forms. Therefore, 32 women with RA were finally included in the intervention group. In the control group, 40 patients were interviewed at baseline. In the 3rd month (last interview), seven patients were excluded for the following reasons: four patients did not wish to continue the study and three patients could not be reached. Therefore, 34 women with RA were finally included in the control group. The study included a total of 66 women with RA, including intervention (n= 32) and control (n= 34) groups. Flow chart of data collection for women with RA is presented Figure 1.

Data collection tools Data were collected by The Patient Information Form, Rheumatoid Arthritis Quality of Life Scale, the Health Assessment Questionnaire, and the Hospital Anxiety Depression Scale.

Patient Information Form: Our study was developed by researchers in line with a literature review on the subject. (Bozbas & Gurer, 2018; Fall et al., 2013; Moghadam et al., 2018; Neto et al., 2009). The form consisted of eight questions about sociodemographic characteristics (age, marital status, education, etc.), clinical diagnosis, treatment of RA, concomitant chronic disease, and deformity affected by arthritis.

Rheumatoid Arthritis Patient Education Booklet: The content of the booklet was prepared by researchers in line with the literature. (arthritis.org; Moghadam et al., 2018; nras.org.uk; Rahim & Cheng, 2018). The education topics included description, symptoms, and signs of RA, diagnostic methods, treatment choices, information on medications, RA in pregnancy, disease management information, nutritional recommendations, emotional health, and support in daily living.

Data collection Patients were interviewed twice, at baseline and at the 3rd month. All forms were applied to the patients in the intervention and control groups at baseline. The patients were assigned to the intervention group at random and participated in a one-to-one training program consisting of a 30-min onset session. The Rheumatoid Arthritis Patient Education Booklet prepared by the researchers was administered to patients in the intervention group during education. The inpatients were given one-to-one training in the patient's room during quiet periods. The outpatients were trained in the outpatient clinic, as tis was considered a suitable venue. In the 3rd month, all forms were applied again to the patients in the intervention group, and the same forms were applied to the untrained patients in the control group. The application of the forms took approximately 15 min, and the interviews were conducted face-to-face with the patients.

Data analysis Data were analyzed using IBM SPSS 20.0 program. Socio-demographic data were analyzed using the mean, standard deviation, and frequency. The Mann-Whitney U paired-group test was used to compare results that did not show a normal distribution. The Fisher's exact test, Pearson chi-square test, and continuity correction test were used. The Wilcoxon signed-rank test was used for the paired comparisons in the comparison of qualitative data. The significance level was set at p < 0.05.

Ethical considerations A University Research Ethics Committee was confirmed the study protocol, which adhered to the Helsinki Declaration (Approval number: 2018/344). Before taking part in the study, all of the patients signed consent forms. Participants were informed that their personal information and privacy would be protected. Patients who did not want to continue to participate in the study were free to leave the study at any stage.

ELIGIBILITY:
Inclusion Criteria:

* To be female
* 18 years of age and older
* Diagnosed with Rheumatoid Arthritis who reached the 2010 American College of Rheumatology (ACR) criterion
* Had a disease period of at least 6 months

Exclusion Criteria:

* Other serious and chronic mental disorders
* Communication difficulties
* Illiteracy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The prevalence of Rheumatoid Arthritis prevalence is three times higher in women than in men.
Enrollment: 66 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline Rheumatoid Arthritis Quality of Life Questionnaire in the third month | Patients' quality of life assess at baseline and in the third month.
  The questionnaire consists of 30 questions, each with a score of "yes" = 1 or "no" = 0. The scores ranged from 0 to 30, with high scores showing poor quality of life.

SECONDARY OUTCOMES:
Change from baseline Hospital Anxiety and Depression Scale (HADS) in the third month | Patients' HADS scores assess at baseline and in the third month.
  The HADS includes both anxiety and depression subscales, and consists of 14 items, 7 of which examine depression and 7 of which examine anxiety. Answers are assessed on a four-point likert scale and graded between 0 and 3. The purpose of the scale is not to diagnose but to assess the risk group by checking for anxiety and depression over a short period
Change from baseline Stanford Health Assessment Questionnaire (HAQ) in the third month | Patients' HAQ score assess at baseline and the third month.
  The HAQ is composed of 20 questions that are divided into eight categories: waking up, moving, feeding, dressing and grooming, hygiene, grip, reach, and tasks. Every question has four possible answers: no challenge (0), some difficulty (1), a lot of difficulty (2), and unable to do (3). the score is computed as an average of eight domains with scores varying from 0 to 3, with a higher score displayed significant impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Irem Yildiz Cilengiroglu, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No